CLINICAL TRIAL: NCT01378793
Title: Acupressure for Chronic Insomnia in Adults With Chronic Low Back Pain
Brief Title: Acupressure for Insomnia
Acronym: AcuSnooze
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollement
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Suzanna Zick, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OVPR-235500
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Insomnia
Keywords: Acupressure; Insomnia; Sleep Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care (No Intervention): Participants will be asked to continue doing whatever their healthcare providers advise for their insomnia, but not to start any new treatments during the study. They will also be given a sleep hygiene handout as a standard of care. After six weeks, they will be reassessed and then provided the opportunity to engage in the web-based acupressure intervention.
- Relaxation Acupressure (Active Comparator): In addition to being given a sleep hygiene handout as a standard of care, participants will be asked to apply pressure on each of following points (bilaterally where indicated). There are 5 acupoints with 4 of the acupoints performed on both the left and the right sides of the body giving a total of 9 points to stimulate. Each of the 9 acupoints will be stimulated for 3 minutes per point giving a total treatment time of 27 minutes done once daily.
  Interventions: Behavioral: Relaxation Acupressure
- Stimulating Acupressure (Active Comparator): In addition to being given a sleep hygiene handout as a standard of care, participants will be asked to apply pressure on each of following points (bilaterally where indicated). There are 6 acupoints with 4 of the acupoints performed on both the left and the right sides of the body giving a total of 10 points to stimulate. Each of the 10 acupoints will be stimulated for 3 minutes per point giving a total treatment time of 30 minutes done once daily.
  Interventions: Behavioral: Stimulating Acupressure

INTERVENTIONS:
Behavioral: Relaxation Acupressure — Apply pressure (stimulate) to the 9 acupoints for 3 minutes per point giving a total treatment time of 27 minutes done once daily for a period of 6 weeks.
  Arms: Relaxation Acupressure
Behavioral: Stimulating Acupressure — Apply pressure (stimulate) to the 10 excitatory acupoints for 3 minutes per point giving a total treatment time of 30 minutes done once daily for a period of 6 weeks.
  Arms: Stimulating Acupressure

SUMMARY:
The purpose of this study is to examine the effect of 6-weeks of relaxation acupressure compared to stimulating acupressure or a standard of care on sleep and daytime functioning. Also, to evaluate the ability of teaching acupressure using web-based applications.

It is believed that self-administered relaxation acupressure will result in improvements of sleep quality and quantity as compared to stimulating acupressure or a standard of care.

DETAILED DESCRIPTION:
Insomnia is a significant health problem and is associated with increased mental health issues: It is estimated that 9% to 15% of the adult population suffers from chronic insomnia. These estimates are considerably higher in primary care where from 20% to 33% suffer from chronic insomnia. Insomnia adversely affects psychological, physical and occupational functioning and places a significant burden on society. Moreover, several cohort studies have found that people with insomnia have significantly higher absenteeism at work, report poor self-esteem, less job satisfaction, and less efficiency at work compared to good sleepers.

Acupressure is a TCM technique based on a philosophy similar to that of acupuncture (the placement and stimulation of very fine needles into acupuncture points). Acupressure involves placing physical pressure by fingers, thumb, elbow, or with the aid of various devices such as pencil erasers on different acupuncture points (acupoints). Depending on the date of the review and the inclusion criteria, e.g., searched in Chinese language databases, there are anywhere from 7^12 to 4^68 randomized clinical trials (RCT) of various types of acupuncture (inclusive of acupressure) for treating insomnia. Regardless of the review the conclusions are remarkably consistent. Mainly, that the majority of RCTs demonstrated that acupuncture was significantly more effective than BDZs, sleep hygiene counseling, no treatment and sham acupuncture for treating insomnia.

The investigators will attempt to prove that self-administered Relaxation Acupressure (RA) will result in improvements in measures of sleep quality and quantity, compared to Stimulating Acupressure (SA) and a wait list control (WL). Also, that they will be able to teach the acupressure points using a web-based application.

Participants will be randomized into 1 of 3 arms; RA, SA, or WL (standard of care). If randomized into one of the acupressure arms, the participants will view their appropriate acupressure training lesson online and be tested on their understanding. They will also be asked to perform their acupoints once per day for a total of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Meet DSM-IV criteria for primary insomnia
* Insomnia must also be documented on two weeks of a baseline sleep diary

Exclusion Criteria:

* Diagnosis or high clinical suspicion of a sleep disorder other than insomnia
* Evidence of a unstable Axis I psychiatric disorder
* Evidence of an uncontrolled medical disorder or pain syndrome that affects sleep, causes daytime sleepiness, or is likely to be causally associated with the insomnia
* Current pharmacological or non-pharmacological insomnia treatment
* Routine overnight shift work
* Previous failed trial of acupuncture or acupressure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-06-15 (Actual); Primary Completion 2013-12-15 (Actual); Study Completion 2013-12-15 (Actual)

PRIMARY OUTCOMES:
Difference in the effect of 6-weeks of Relaxation Acupressure compared to Stimulating Acupressure or standard of care on chronic insomnia and daytime functioning. | 6 weeks
  Insomnia will be assessed/determined by daily sleep/wake diaries and the Insomnia Severity Index questionnaire. Sleep Diary: insomnia = <85% sleep efficiency ratio.
  Daytime functioning will be determined by the Fatigue Severity Scale of Sleep Disorders (FSS).

SECONDARY OUTCOMES:
Success of teaching the acupressure interventions using a novel web-based application measured by an Acupressure Fidelity Form at week 1 and week 6. | 6 weeks
  The success of learning acupressure via a web-based application will be assessed using an Acupressure Fidelity Form. The form will assess the participants ability to locate each acupressure point, demonstrate proper pressure/technique, and know the frequency of their treatments. Acupressure Form A is worth a total of 12 points while Form B is worth 13 points. Each correct answer is worth 1 point. We will consider our web based intervention "successful" if 95% of participants (49 of them) received a score of 100% at both visits.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Zick, ND, MPH, Principal Investigator — , Department of Family Medicine, University of Michigan; Richard E Harris, PhD, Principal Investigator — , Departments of Anesthesiology and Internal Medicine, University of Michigan
Locations (1):
- Domino's Farm, Ann Arbor, Michigan, United States